CLINICAL TRIAL: NCT05847426
Title: Improving Early Intervention in Hearing Impaired Children Using Functional Near-Infrared Spectroscopy (fNIRS)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Bionics Institute of Australia (Other)
Responsible Party: Principal Investigator, Colette McKay, Leader, Translational Hearing Research and Principal Scientist, The Bionics Institute of Australia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 90457
Record Dates: First submitted 2023-04-27; First posted 2023-05-06 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Hearing Impairment
Keywords: Infants; Early intervention; functional near-infrared spectroscopy
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Intervention Model Description: The intervention (provision of additional fNIRS information) will be applied to audiologists in a cross-over design, wherein each audiologist will receive the anonymized current audiological information about a particular infant twice: once with, and once without the additional fNIRS information. Each time, the audiologist will answer questions about key management decisions via a questionnaire and rate their confidence in their decision using a sliding scale. The change in confidence (difference between the two sliding scale answers for the audiologist) when having access to additional fNIRS information will be the raw data analysed.
  To test the main hypothesis (that including fNIRS information increases confidence in making management decisions) separately for different hearing loss category groups and different points in the care pathway, 232 infants will be recruited to undergo fNIRS testing, divided into subgroups each with target numbers based on power calculation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Provision of standard audiological + fNIRS test results (Experimental): The treatment arm involves the provision of additional fNIRS sound detection and speech discrimination test results to the audiologists, in addition to standard audiology information. Standard information includes:
  1. At diagnosis: unaided Auditory Brainstem Response results;
  2. After initial hearing aid provision: as a) above plus aided Cortical Evoked Potentials;
  3. After hearing aid program is adjusted to satisfaction: as b) above plus parent observational report, PEACH (2);
  4. After initial cochlear implant programming: behavioural observations.
  Interventions: Other: Provision of standard audiological + fNIRS test results
- Provision of standard audiological test results only (Active Comparator): The standard audiology information available to the audiologists includes:
  1. At diagnosis: unaided Auditory Brainstem Response results;
  2. After initial hearing aid provision: as a) above plus aided Cortical Evoked Potentials;
  3. After hearing aid program is adjusted to satisfaction: as b) above plus parent observational report, PEACH (2);
  4. After initial cochlear implant programming: behavioural observations.
  Interventions: Other: Provision of standard audiological test results only

INTERVENTIONS:
Other: Provision of standard audiological + fNIRS test results — Infants with hearing loss will be tested using functional near-infrared spectroscopy (fNIRS) and a patented analysis algorithm to measure sound detection and discrimination. Their standard audiological test results will also be collected from their audiology service provider/s. Both sets of test results will be given to the participating audiologists in the experimental arm.
  Arms: Provision of standard audiological + fNIRS test results
Other: Provision of standard audiological test results only — The provision of test results to the audiologist will be the same as in the experimental arm, but without the fNIRS test results included.
  Arms: Provision of standard audiological test results only

SUMMARY:
The goal of this clinical trial is to find out whether hearing test results using functional near-infrared spectroscopy (fNIRS) will help to fast-track early intervention for infants born with a hearing loss. fNIRS is a method of imaging brain activity using light. The main questions are:

1. Can audiologists make more confident decisions about the optimal interventions at different critical points in the hearing care pathway when they are given additional fNIRS information compared to when they have standard audiology test results alone?
2. Is the experience of their infant having an fNIRS test acceptable and comfortable for the parents or care givers?

DETAILED DESCRIPTION:
Universal newborn hearing screening (UNHS) has reduced the age of diagnosis of permanent childhood hearing loss from several years down to several weeks. While this is highly desirable, the early diagnosis raises challenges for the audiologists who manage these infants. The challenges are due to a lack of relevant audiological information, particularly about an infant's ability to discriminate between different speech sounds, and, for infants with Auditory Neuropathy, their degree of hearing impairment, which is required to make key management decisions. The missing information causes intervention delays at several time-critical points along the standard hearing care pathway that could seriously affect speech and language development for the infant, with life-long social, educational and employment consequences. The goal of this trial is to assess whether the addition of audiological information provided by fNIRS assessments can address these challenges for audiologists who care for infants with different types of hearing loss and at the different critical decision points in the care pathway.

A pool of at least 40 experienced audiologists will be recruited to participate in the study. In addition, infants with different types and degree of hearing loss, and at the different critical points in their care pathway will be recruited to provide fNIRS test results. For each infant, a group of ten paediatric audiologists will be randomly selected from the large pool and will be provided with anonymised audiological test results. Each audiologist will receive the current test results of the infant twice, once with, and once without the additional fNIRS test results, with 2 months between. Half (5 randomly selected) will receive the standard plus additional fNIRS test results before the standard-alone results and the other half in reverse order. The audiologists will be asked, via a questionnaire, to make clinical decisions relevant to the infant's point in the hearing care pathway and to rate their confidence in their decisions on a sliding scale.

Infants will be recruited for fNIRS tests at each of four points in the care pathway (after diagnosis, after first hearing aid provision, when optimal hearing aid program is established, and after cochlear implantation. The critical management decisions at these four points are, respectively: Is a hearing aid needed?; Is the hearing aid optimally programmed for the infant?; Would the infant be better off with a cochlear implant instead of their hearing aid?; and Is the cochlear implant programmed optimally for the infant?

Parents/guardians will also be surveyed about their experience with the fNIRS test.

ELIGIBILITY:
The above eligibility applies to the participating audiologists who are in the experimental and control arms of the study

Audiologist Inclusion Criteria:

* Is a qualified audiologist who meets the criteria for membership of Audiology Australia.
* Has at least 1 year of experience in paediatric diagnostic, hearing aid or cochlear implant audiology service provision in Australia.
* Provides a signed and dated informed consent form.

Audiologist Exclusion criteria (only for a specific infant test result):

* Is the managing audiologist for the infant who's results are being provided.

Infants are also recruited into the study to have an fNIRS assessment performed. They do not participate further after the fNIRS test.

Infant Inclusion criteria:

* Between the ages of 1 and 24 months at the time of fNIRS testing.
* Has permanent hearing loss in one or both ears as determined by audiological diagnostic testing.
* Has a legally acceptable representative capable of understanding the informed consent document and providing consent on the participant's behalf.

Infant Exclusion Criteria:

* There are no exclusion criteria other than not meeting the inclusion criteria.

Min Age: 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-05-02 (Actual); Primary Completion 2028-04-28 (Estimated); Study Completion 2028-04-28 (Estimated)

PRIMARY OUTCOMES:
Change in confidence of audiological clinical management decisions when fNIRS hearing test results are included with standard audiological information compared to when using standard information alone | Between each infant's completed fNIRS testing session and 2 months after
  The questionnaire responses that the participating audiologists provide will measure their confidence in making the appropriate next decision for the infant using a sliding scale (0 (no confidence) to 100 (high confidence)). The data from the sliding scale responses for the same audiologist/infant will be subtracted (confidence with fNIRS minus confidence without fNIRS) to obtain the raw data for analysis.

SECONDARY OUTCOMES:
Parental/Guardian perception of acceptability of fNIRS test process and usefulness of fNIRS test results | Within 2 weeks after their child's fNIRS testing session
  The results of a parent questionnaire developed by the Advisory Committee (which includes parent members) will be qualitatively evaluated to determine if the fNIRS test process was acceptable, and the test results were perceived as useful. The results will also indicate whether there are aspects of the test process that could be improved in future to make it more acceptable to parents.

CONTACTS AND LOCATIONS:
Overall Officials: Professor Colette McKay, Principal Investigator — The Bionics Institute of Australia
Locations (5):
- Australia (5):
  - The Royal Victorian Eye and Ear Hospital, East Melbourne, Victoria
  - Bionics Institute, Fitzroy, Victoria
  - Barwon Health, Geelong, Victoria
  - Hearing Australia, Moonee Ponds, Victoria
  - The Royal Children's Hospital, Parkville, Victoria

IPD SHARING:
Plan to Share IPD: Yes
Beginning 1 month following analysis and article publication, the following data will be made available long-term for use by future researchers from a recognised research institution whose proposed use of the data has been ethically reviewed and approved by an independent committee and who accept Bionics Institute's conditions for access:
  * Raw anonymized confidence rating scores linked to the questionnaire question, infant subgroup (type and degree of hearing loss categories), and point in clinical care pathway.
  * study protocol and statistical analysis plan if not already clear in the publication
Supporting Information: Study Protocol, SAP
Time Frame: Data, study protocol, and statistical analysis plan will be available from one month following trial analysis and article publication, for a period of 10 years.
Access Criteria: Data can only be accessed if the researchers are from a recognized research institution, the proposed use of the data has been ethically reviewed and approved by an independent committee, and the researchers accept Bionics Institute's conditions for access.

REFERENCES:
- [Background] Mao D, Wunderlich J, Savkovic B, Jeffreys E, Nicholls N, Lee OW, Eager M, McKay CM. Speech token detection and discrimination in individual infants using functional near-infrared spectroscopy. Sci Rep. 2021 Dec 14;11(1):24006. doi: 10.1038/s41598-021-03595-z. PMID 34907273
- [Background] Paranawithana I, Mao D, Wong YT, McKay CM. Reducing false discoveries in resting-state functional connectivity using short channel correction: an fNIRS study. Neurophotonics. 2022 Jan;9(1):015001. doi: 10.1117/1.NPh.9.1.015001. Epub 2022 Jan 18. PMID 35071689
- [Background] Shader MJ, Luke R, Gouailhardou N, McKay CM. The use of broad vs restricted regions of interest in functional near-infrared spectroscopy for measuring cortical activation to auditory-only and visual-only speech. Hear Res. 2021 Jul;406:108256. doi: 10.1016/j.heares.2021.108256. Epub 2021 Apr 28. PMID 34051607
- [Background] Zhou X, Sobczak G, McKay CM, Litovsky RY. Comparing fNIRS signal qualities between approaches with and without short channels. PLoS One. 2020 Dec 23;15(12):e0244186. doi: 10.1371/journal.pone.0244186. eCollection 2020. PMID 33362260
- [Background] Weder S, Shoushtarian M, Olivares V, Zhou X, Innes-Brown H, McKay C. Cortical fNIRS Responses Can Be Better Explained by Loudness Percept than Sound Intensity. Ear Hear. 2020 Sep/Oct;41(5):1187-1195. doi: 10.1097/AUD.0000000000000836. PMID 31985534
- [Background] Weder S, Zhou X, Shoushtarian M, Innes-Brown H, McKay C. Cortical Processing Related to Intensity of a Modulated Noise Stimulus-a Functional Near-Infrared Study. J Assoc Res Otolaryngol. 2018 Jun;19(3):273-286. doi: 10.1007/s10162-018-0661-0. Epub 2018 Apr 9. PMID 29633049